CLINICAL TRIAL: NCT01827943
Title: Phase II Trial, Evaluating Efficacy of Temsirolimus (Torisel ®) in Second Line Therapy for Patients With Advanced Bladder Cancer
Brief Title: Phase II Evaluating Efficacy of Temsirolimus in 2 Line Therapy for Patients With Advanced Bladder Cancer
Acronym: VESTOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2009-08
Record Dates: First submitted 2012-10-29; First posted 2013-04-10 (Estimated); Results first posted 2021-04-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Relapsed Bladder Cancer
Keywords: Relapsed bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus (Experimental): Temsirolimus was administered intravenously at a dose of 25 mg in a weekly 30 min infusion and was associated to anti-H1 treatment. One cycle corresponded to 4 weeks of treatment.
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — Temsirolimus
  Other Names: Torisel

SUMMARY:
In the absence of standard treatment in this indication, this test evaluates a new drug type targeted therapy in this indication, evaluating its efficacy in terms of tumor response and survival.

DETAILED DESCRIPTION:
In the absence of standard treatment in this indication, this test evaluates a new drug type targeted therapy in this indication, evaluating its efficacy in terms of tumor response and survival. This study will also search for genes involved in the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of at least 18 years of age
* Histologically proven Bladder cancer
* Locally advanced or metastatic disease (stage IV)
* Functional status (ECOG / OMS) ≤ 2
* Relapse after first-line chemotherapy
* Measurable lesions (RECIST criteria)
* Absence of anti-neoplasic treatment in the 4 weeks preceding inclusion.
* Biological levels :
* Neutrophil count >1,5.109/L.
* Platelets >100.109/L
* Total serum bilirubin < 1.5 × ULN
* Clearance of créatinine 40 ml/mm
* If not liver metastasis alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 × ULN
* With liver alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <5 × ULN
* Signed informed consent
* Both women and men must agree to use a medically acceptable method of contraception throughout the study. Women of childbearing potential must have a negative serum pregnancy test of or less than 7 days before the first perfusion of study.
* France only : Patients affiliated to a social security program

Exclusion Criteria:

* Presence of metastatic brain or meningeal tumors on selection scanner, weither symptomatic or asymptomatic
* Chemotherapy, immunotherapy, or radiotherapy within 4 weeks of inclusion
* Known hypersensitivity to temsirolimus, or its metabolites (as sirolimus), or polysorbate 80 or to their excipients
* Previous malignancy (except for cervical carcinoma in situ, basal cell carcinoma curatively treated) or incidental (≤ pT2) prostate cancer found on a radical cystoprostatectomy material
* The drugs known as CYP3A4/5 inhibitors or inducers will specifically be excluded on the 30th day ( or at least 7 halves-lives, according to the shortest duration) before the first perfusion and throughout the study. Any food known to inhibit CYP3A4/5 (for example grapefruit, grapefruit juice, star-fruit or star-fruit juice) will also be purposely excluded.
* Auto-immune pathology, psychiatric or neurological disorder
* Any unstable medical condition
* Unstable cardiac disease
* Severe renal failure
* Unstable diabetes
* Pregnancy
* Patient enrolled in another therapeutic clinical trial
* Patient unable to follow and comply with the study procedures because of any geographical, social or medical condition
* Patient partially or totally deprived of his civil rights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-06; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine HOUEDE, MD, Study Chair — Institut Bergonié
Locations (9):
- France (9):
  - CHU de Bordeaux, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - Centre Léon Bérard, Lyon
  - Hôpital d'instruction des armées du Val-de-Grâce, Paris
  - CHU de Rouen, Rouen
  - Institut Claudius Regaud, Toulouse
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Result] Pulido M, Roubaud G, Cazeau AL, Mahammedi H, Vedrine L, Joly F, Mourey L, Pfister C, Goberna A, Lortal B, Bellera C, Pourquier P, Houede N. Safety and efficacy of temsirolimus as second line treatment for patients with recurrent bladder cancer. BMC Cancer. 2018 Feb 17;18(1):194. doi: 10.1186/s12885-018-4059-5. PMID 29454321

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temsirolimus
Started | 54
Safety Population (Safety population included patients with at least one administration of treatment) | 53
Completed | 45
Not Completed | 9
Not completed — Protocol Violation | 8
Not completed — Never treated because of an rapid progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Temsirolimus
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 65.0 [41.0 to 87.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Non-progression Rate at 2 Months
Description: Non-progression rate is defined as the rate of participants in complete or partial response or stable disease according to RECIST V1.1.
  Complete response is defined as the disappearance of all target lesions, partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters and stable disease occurs when neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progression, taking as reference the smallest sum diameters while on study.
Time Frame: 2 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temsirolimus
Number analyzed (Participants) | 45
percentage of participants | 48.9 [33.7 to 64.2]

2. Secondary Outcome: Overall Survival
Description: OS was was defined as the time from the treatment initiation to death due to any cause. Participants without documented death were censored at the date of the last follow-up or last patient contact. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Through Database Cutoff Date of 23-Jan-2015 (up to approximately 5 years and 7 months - median follow-up time of 14 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus
Number analyzed (Participants) | 45
months | 7.2 [5.2 to 9.5]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from the initiation of treatment to the first documented progression (as per RECIST v1.1) or death (due to any cause), whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Patients alive and progression free were censored at the date of last follow-up or last patient contact. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus
Number analyzed (Participants) | 45
months | 2.8 [1.8 to 3.7]

ADVERSE EVENTS:
Arm/Group | Temsirolimus
All-Cause Mortality (participants affected / at risk) | 40/53
Serious Adverse Events (participants affected / at risk) | 35/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus (N=53)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3) — Blood/Bone Marrow (SOC from CTCAE v3.0)
Platelets (Investigations) | 3 (3) — Blood/Bone Marrow (SOC from CTCAE v3.0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 6 (7) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 13 (15) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1) — GASTROINTESTINAL (SOC from CTCAE v3.0)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 2 (2) — GASTROINTESTINAL (SOC from CTCAE v3.0)
Obstruction, GI (Gastrointestinal disorders) | 4 (5) — GASTROINTESTINAL (SOC from CTCAE v3.0)
Vomiting (Gastrointestinal disorders) | 1 (1) — GASTROINTESTINAL (SOC from CTCAE v3.0)
Hemorrhage, CNS (Nervous system disorders) | 2 (2) — HEMORRHAGE/BLEEDING (SOC from CTCAE v3.0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1) — HEPATOBILIARY / PANCREAS (SOC from CTCAE v3.0)
Infection - Other (Specify, __) (Infections and infestations) | 9 (10) — INFECTION (SOC from CTCAE v3.0)
Infection with unknown ANC (Infections and infestations) | 1 (1) — INFECTION (SOC from CTCAE v3.0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) — METABOLIC LABORATORY (SOC from CTCAE v3.0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) — MUSCULOSKELETAL/SOFT TISSUE (SOC from CTCAE v3.0)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1 (1) — MUSCULOSKELETAL/SOFT TISSUE (SOC from CTCAE v3.0)
Confusion (Psychiatric disorders) | 1 (1) — NEUROLOGY (SOC from CTCAE v3.0)
Mood alteration (Psychiatric disorders) | 1 (1) — NEUROLOGY (SOC from CTCAE v3.0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — PAIN (SOC from CTCAE v3.0)
Pain - Other (Specify, __) (General disorders) | 5 (7) — PAIN (SOC from CTCAE v3.0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — PULMONARY / UPPER RESPIRATORY (SOC from CTCAE v3.0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 3 (3) — PULMONARY / UPPER RESPIRATORY (SOC from CTCAE v3.0)
Renal failure (Renal and urinary disorders) | 2 (2) — RENAL/GENITOURINARY (SOC from CTCAE v3.0)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 2 (2) — RENAL/GENITOURINARY (SOC from CTCAE v3.0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) — RENAL/GENITOURINARY (SOC from CTCAE v3.0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus (N=53)
Hemoglobin (Blood and lymphatic system disorders) | 26 (40) — Blood/Bone Marrow (SOC from CTCAE v3.0)
Leukocytes (total WBC) (Investigations) | 3 (4) — Blood/Bone Marrow (SOC from CTCAE v3.0)
Platelets (Investigations) | 16 (24) — Blood/Bone Marrow (SOC from CTCAE v3.0)
Hypertension (Vascular disorders) | 4 (4) — CARDIAC GENERAL (SOC from CTCAE V3.0)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 20 (21) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 39 (43) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 21 (26) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Insomnia (Psychiatric disorders) | 5 (5) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Weight loss (Investigations) | 11 (12) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 13 (20) — DERMATOLOGY/SKIN (SOC from CTCAE V3.0)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (14) — DERMATOLOGY/SKIN (SOC from CTCAE V3.0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8 (11) — DERMATOLOGY/SKIN (SOC from CTCAE V3.0)
Rash/desquamation (Injury, poisoning and procedural complications) | 8 (10) — DERMATOLOGY/SKIN (SOC from CTCAE V3.0)
Anorexia (Metabolism and nutrition disorders) | 23 (26) — Gastrointestinal (SOC from CTCAE V3.0)
Constipation (Gastrointestinal disorders) | 13 (13) — Gastrointestinal (SOC from CTCAE V3.0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) — Gastrointestinal (SOC from CTCAE V3.0)
Diarrhea (Gastrointestinal disorders) | 15 (20) — Gastrointestinal (SOC from CTCAE V3.0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (3) — Gastrointestinal (SOC from CTCAE V3.0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 3 (3) — Gastrointestinal (SOC from CTCAE V3.0)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 3 (3) — Gastrointestinal (SOC from CTCAE V3.0)
Hemorrhoids (Gastrointestinal disorders) | 3 (5) — Gastrointestinal (SOC from CTCAE V3.0)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 19 (23) — Gastrointestinal (SOC from CTCAE V3.0)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 3 (4) — Gastrointestinal (SOC from CTCAE V3.0)
Nausea (Gastrointestinal disorders) | 23 (24) — Gastrointestinal (SOC from CTCAE V3.0)
Obstruction, GI (Gastrointestinal disorders) | 6 (7) — Gastrointestinal (SOC from CTCAE V3.0)
Taste alteration (dysgeusia) (Nervous system disorders) | 10 (10) — Gastrointestinal (SOC from CTCAE V3.0)
Vomiting (Gastrointestinal disorders) | 15 (19) — Gastrointestinal (SOC from CTCAE V3.0)
Hemorrhage, GU (Renal and urinary disorders) | 3 (5) — HEMORRHAGE/BLEEDING (SC from CTCAE V3.0)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 6 (6) — HEMORRHAGE/BLEEDING (SC from CTCAE V3.0)
Infection - Other (Specify, __) (Infections and infestations) | 31 (45) — INFECTION (SOC from CTCAE V3.0)
Edema:limb (General disorders) | 14 (14) — LYMPHATICS (SOC from CTCAE V3.0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (3) — METABOLIC/LABORATORY (SOC from CTCAE V3.0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (4) — METABOLIC/LABORATORY (SOC from CTCAE V3.0)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 7 (7) — METABOLIC/LABORATORY (SOC from CTCAE V3.0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (6) — METABOLIC/LABORATORY (SOC from CTCAE V3.0)
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 3 (3) — METABOLIC/LABORATORY (SOC from CTCAE V3.0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3) — METABOLIC/LABORATORY (SOC from CTCAE V3.0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (6) — METABOLIC/LABORATORY (SOC from CTCAE V3.0)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 13 (16) — METABOLIC/LABORATORY (SOC from CTCAE V3.0)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 6 (6) — MUSCULOSKELETAL/SOFT TISSUE (SOC from CTCAE V3.0)
Dizziness (Nervous system disorders) | 3 (3) — NEUROLOGY (SOC from CTCAE V3.0)
Mood alteration (Psychiatric disorders) | 13 (15) — NEUROLOGY (SOC from CTCAE V3.0)
Neuropathy: sensory (Nervous system disorders) | 6 (8) — NEUROLOGY (SOC from CTCAE V3.0)
Pain (General disorders) | 29 (61) — PAIN (SOC from CTCAEV3.0)
Pain - Other (Specify, __) (General disorders) | 5 (6) — PAIN (SOC from CTCAEV3.0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) — PULMONARY/UPPER RESPIRATORY (SOC from CTCAE V3.0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (7) — PULMONARY/UPPER RESPIRATORY (SOC from CTCAE V3.0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 4 (4) — PULMONARY/UPPER RESPIRATORY (SOC from CTCAE V3.0)
Renal failure (Renal and urinary disorders) | 9 (10) — RENAL/GENITOURINARY (SOC from CTCAE V3.0)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 4 (4) — RENAL/GENITOURINARY (SOC from CTCAE V3.0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes